CLINICAL TRIAL: NCT01378832
Title: Effect of Peritoneal Lavage With Clindamycin-gentamicin Solution on Infection in Elective Surgery
Brief Title: Effect of Peritoneal Lavage With Clindamycin-gentamicin Solution on Postoperative Colorectal Cancer Infection in Elective Surgery
Acronym: lavage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Jaime Ruiz-Tovar, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: jruiztovar
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2010-01

CONDITIONS: Surgical Site Infection
Keywords: Intra-abdominal abscess; wound infection; colorectal surgery
MeSH Terms: conditions — Surgical Wound Infection; Abdominal Abscess; Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Intra-peritoneal antibiotic lavage — The lavage was performed immediately prior to closure of the abdominal wall. Prior to the lavage, a microbiological sample from the peritoneal surface (parietal and visceral) was obtained with a swab (sample 1), followed by a lavage with 500 ml normal saline, similar to the one performed in Group 1. After this lavage, a new microbiological sample was obtained from the peritoneal surface (sample 2), and a second lavage with an antibiotic solution, including gentamicin (240 mg) and clindamycin (600 mg) dissolved in 500 ml normal saline was performed. During this lavage, the solution was allowed to sit in the abdominal cavity for 3 minutes. After aspirating the lavage, a third microbiological sample was obtained in the same way as the two previous ones (sample 3).

SUMMARY:
Intrabdominal antibiotic irrigation will reduce wound and intrabdominal infection.

DETAILED DESCRIPTION:
A prospective, randomized study was performed between January and December 2010. Patient inclusion criteria were a diagnosis of colorectal neoplasms and plans to undergo an elective curative surgery. Patients were divided into 2 groups: Group 1 (intra-abdominal irrigation with normal saline) and Group 2 (intraperitoneal irrigation with a solution of 240 mg gentamicin and 600 mg clindamycin). The occurrence of wound infections and intra-abdominal abscesses were investigated. Following the anastomosis, a microbiological sample of the peritoneal surface was obtained (sample 1). A second sample was collected following an irrigation with normal saline (sample 2). Finally, the peritoneal cavity was irrigated with a gentamicin-clindamycin solution and a third sample was obtained (sample 3).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of colorectal neoplasms and plans to undergo an elective surgery with curative aims.

Exclusion Criteria:

* preoperative diagnosis of chronic renal failure, because of the risk of nephrotoxicity associated with intraperitoneal gentamicin absorption
* an anastomotic leak in the postoperative course

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30 days
  Intra-abdominal abscess and wound infection will be investigated during the first 30 days after colorectal surgery

REFERENCES:
- [Derived] Ruiz-Tovar J, Santos J, Arroyo A, Llavero C, Armananzas L, Lopez-Delgado A, Frangi A, Alcaide MJ, Candela F, Calpena R. Effect of peritoneal lavage with clindamycin-gentamicin solution on infections after elective colorectal cancer surgery. J Am Coll Surg. 2012 Feb;214(2):202-7. doi: 10.1016/j.jamcollsurg.2011.10.014. PMID 22265220